CLINICAL TRIAL: NCT02918578
Title: Tailored Multicomponent Intervention for Remote Physical Activity Promotion in Inactive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Xenia Fischer, M.Sc., University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-00560
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Sedentary Lifestyle
Keywords: Physical Inactivity; Behavior Change
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- "Phone" group (Experimental): see intervention description
  Interventions: Other: "Phone" group
- "Phone and SMS" group (Experimental): see intervention description
  Interventions: Other: "Phone and SMS" group
- "single writing" group (Active Comparator): see intervention description
  Interventions: Other: "single writing" group

INTERVENTIONS:
Other: "Phone" group — Participants in the "phone" group receive 12 individually tailored coaching sessions (15 - 20 min). The coaching calls are scheduled biweekly. Participants receive their tailored advice via interactive counseling.
  Arms: "Phone" group
Other: "Phone and SMS" group — The "phone and SMS" group receive the same coaching as the "phone" group. They additionally receive two tailored SMS per week over the course of six months.
  Arms: "Phone and SMS" group
Other: "single writing" group — The control intervention consists of a "minimal credible" physical activity PA promotion program. Participants in the control group receive a singular written advice and an activity plan but no counseling by phone.
  Arms: "single writing" group

SUMMARY:
The purpose of this study is to compare different modalities to communicate a remote and individually tailored physical activity promotion program.

DETAILED DESCRIPTION:
Physical inactivity (PI) adversely affects various non-communicable diseases (WHO, 2010) and has been recently entitled "the biggest public health problem of the 21th century" (Blair, 2009). Despite the strong evidence for physical activity (PA) related health benefits, one third of the world's population is physically inactive (Hallal et al., 2012). In Switzerland, 35% of the adults are not meeting the minimum recommendation of 2.5h moderate to vigorous activity per week (BASPO, 2013). Present PI patters accompanied with demographic changes and the burden of non-communicable diseases (WHO, 2010) constitute a notable challenge to the health-care system. Thus, effective prevention programs that engage individuals to become more physically active are needed and of public interest.

Regarding the application for a wide public, the use of technologies for a remote delivery of PA promotion programs is promising (Castro & King, 2002). Thereby, PA lifestyle interventions including individually tailored program components (Noar, Benac, & Harris, 2007), personal coaching (Foster, Richards, Thorogood, & Hillsdon, 2013), behavior change techniques (BCT) (Michie, Abraham, Whittington, McAteer, & Gupta, 2009) and regular prompting (push notifications) (De Leon, Fuentes, & Cohen, 2014) are regarded as effective means to improve PA behavior. However, it is still not examined to date, which intervention components could be effectively translated into practice. The required density, the most effective modality and long-term outcomes of PA promotion program need to be examined (Foster et al., 2013).

Within this study three versions to communicate an individually tailored PA promotion program will be compared. The program consists of individual counseling but is delivered without face-to-face contact. Exercise recommendations and behavior change techniques will be elaborated on an individual basis, communicated and assessed. The programs content will then be tailored according to personal background information (e.g. goals, preferences) assessed by questionnaires.

A personalized activity-profile on a specifically developed internet portal (on www.movingcall.com) enables safe exchange between participant and coach. The activity-profile includes a weekly activity plan, questionnaires and a diary to document daily PA behavior.

All enrolled participants will have access to a personal activity profile and receive a tailored advice to increase their physical activity levels. Depending on the interventional arm the advice will be delivered in a more supportive and interactive manner. Participants will be randomly assigned to one of the three study arms.

The primary objective is to assess the effect of regular coaching and prompting on PA level. Secondary objectives are the assessment of follow-up effects of PA changes and changes in psychosocial determinants of PA as well as the comparison self-reported and objectively assessed PA data.

Outcome measures will be assessed prior to the start of the intervention, at the end of the six months and in the follow-up period after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* not meeting the physical activity guidelines of 150 minutes moderate or 75 minutes vigorous aerobic activity

Exclusion Criteria:

* medical condition that contraindicates the participation in regular moderate-intensity exercise

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2016-08; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Self-reported physical activity level of one week | 6 months of intervention
  Simple Physical Activity Questionnaire; SIMPAQ
Objectively assessed physical activity level of one week | 6 months of intervention
  Accelerometer

SECONDARY OUTCOMES:
Self-reported physical activity level of one week | In the follow-up after 12 months
  Simple Physical Activity Questionnaire; SIMPAQ
Objectively assessed physical activity level of one week | In the follow-up after 12 months
  Accelerometer
body weight | At baseline, 6 months and in the follow-up after 12 months
health related quality of life (questionnaire) | At baseline, 6 months and in the follow-up after 12 months
  Health related quality of life will be assessed by the Short Form 12 Questionnaire (SF-12) (Bullinger, 1995; Ware, Kosinski, & Keller, 1996). The questionnaire includes 12 items on general physical health status and mental health distress.
stress-related exhaustion symptoms (questionnaire) | At baseline, 6 months and in the follow-up after 12 months
  Perceived stress-related exhaustion symptoms will be measured by the validated Shirom-Melamed Burnout Measure (SMBM) (Shirom & Melamed, 2006).
Adherence to the PA promotion program (count data) | At baseline, 6 months and in the follow-up after 12 months
  Adherence will be calculated by the frequency of logins to the personal profile and the frequency of entering self-monitoring data.
Satisfaction with the program (questionnaire) | At baseline, 6 months and in the follow-up after 12 months
  A self-compiled questionnaire will be used to assess general satisfaction, motivation to continue with the program, comprehensibility of the profile and suggestions for future improvements of the program.
Intention on physical activity participation (questionnaire) | At baseline, 6 months and in the follow-up after 12 months
  Motivational readiness will be assessed according to the stages of change of the Transtheoretical Model (Fuchs, 2007; Marcus, Rakowski, & Rossi, 1992).
Outcome expectations on physical activity participation (questionnaire) | At baseline, 6 months and in the follow-up after 12 months
  Outcome expectancies regarding the physical activity will be assessed with eight items according to Fuchs (1994).
Self-efficacy concerning physical activity participation (questionnaire) | At baseline, 6 months and in the follow-up after 12 months
  Consistent with Fuchs (2008), self-efficacy will be assess by the confidence to begin, to maintain and to restart regular physical activity.
Barriers concerning physical activity participation (questionnaire) | At baseline, 6 months and in the follow-up after 12 months
  Perceived barriers: Participants will be presented a list of 19 potential barriers and asked to indicate how strong each one prevented physical activity (Fuchs, Seelig, Gohner, Burton, & Brown, 2012)
Social support for physical activity participation (questionnaire) | At baseline, 6 months and in the follow-up after 12 months
  Social support will be assessed by 7 items that rate the confidence for support of the social environment (Fuchs, 1997).

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Zahner, Prof. Dr., Study Director — Department of Sport, Exercise and Health
Locations (1):
- University of Basel, Department of Sport, Exercise and Health, Basel, Birsstr. 320B, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer X, Donath L, Zwygart K, Gerber M, Faude O, Zahner L. Coaching and Prompting for Remote Physical Activity Promotion: Study Protocol of a Three-Arm Randomized Controlled Trial (Movingcall). Int J Environ Res Public Health. 2019 Jan 25;16(3):331. doi: 10.3390/ijerph16030331. PMID 30691013